CLINICAL TRIAL: NCT03732469
Title: Administration of Rectal Acetaminophen During Oocyte Retrievals Reduces Post-Operative Opioid Utilization in Fertility Patients
Brief Title: Rectal Acetaminophen Use During Oocyte Retrievals to Reduce Post-Operative Opioid Utilization
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Significant change in our clinic structure prevented continued recruitment of patients to the study
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00037883
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use
Keywords: egg retrieval; oocyte retrieval; opioid dependence; rectal acetaminophen; rectal tylenol; pain; opioid use; opioid abuse
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — Acetaminophen; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl/propofol + acetaminophen (Experimental): In addition to the weight-based intraoperative IV dose of propofol and fentanyl per standard TGH Anesthesiology protocol, one dose of 1300 mg of solid base rectal acetaminophen suppository (2 suppositories) will be administered at the end of oocyte retrieval.
  Interventions: Drug: Acetaminophen; Drug: Fentanyl; Drug: Propofol
- Fentanyl/propofol only (Active Comparator): Participants in this arm will receive the weight-based intraoperative IV dose of propofol and fentanyl per standard TGH Anesthesiology protocol.
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Acetaminophen — Rectal acetaminophen will be administered to the intervention group at the conclusion of the oocyte retrieval.
  Other Names: Tylenol
  Arms: Fentanyl/propofol + acetaminophen
Drug: Fentanyl — Weight-based IV Fentanyl as a part of the standard anesthesia/analgesia induction protocol at Tampa General Hospital
Drug: Propofol — Weight-based IV Propofol as a part of the standard anesthesia/analgesia induction protocol at Tampa General Hospital

SUMMARY:
The primary aim of this study is to evaluate the administration of rectal acetaminophen to current and standard anesthesia and analgesia protocol in oocyte retrievals would reduce postoperative utilization of opioids (Tylenol with codeine) in fertility patients.

DETAILED DESCRIPTION:
As the opioid epidemic shows no sign of abating, this national crisis deserves careful attention from all medical subspecialties. This includes reproductive endocrinology and infertility (REI), where opioids are primarily utilized for intraoperative and postoperative pain management for outpatient procedures such as oocyte retrievals, operative hysteroscopy, and laparoscopic myomectomy. The purpose of this study is to evaluate whether the administration of rectal acetaminophen in addition to the current, standard anesthesia and analgesia protocol in oocyte retrievals can help decrease utilization of prescribed opioid at home following oocyte retrieval. Rectal acetaminophen will be used rather than conventional IV acetaminophen because of the lack of access to IV acetaminophen at the study institution. Rectal acetaminophen is appealing because it is cheap, readily available in most medical centers and there is the potential for increased analgesic benefit due to the proximity to the vaginal and ovarian tissue, as well as the possible benefit from the partial avoidance of hepatic first-pass metabolism. This trial has the potential to provide practice-changing clinical information to the field of REI. The information gained can even translate to other ambulatory procedures and guide clinical practice. The investigators hypothesize that participants given rectal acetaminophen in addition to standard anesthesia/analgesia at the end of their oocyte retrieval will use less amount of prescribed Tylenol with codeine 3 days after discharge from the surgery center compared those receiving standard anesthesia/analgesia for oocyte retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Any female patient undergoing oocyte retrieval by transvaginal ultrasound-guided ovarian puncture

Exclusion Criteria:

* Patients with chronic pain conditions such as fibromyalgia and sickle cell anemia.
* Patient with BMI greater than 40
* Patients that required general endotracheal intubation anesthesia in prior oocyte retrieval
* Patients with documented allergic reaction to acetaminophen
* Patient with contra-indication to the use of acetaminophen (liver disease)
* Patients with a history of past or current alcohol, drug or opioid abuse
* Patients with ulcerative colitis, Crohn's disease, or severe rectal hemorrhoids

Ages: 18 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of prescribed Tylenol with Codeine (Tylenol #3) utilized | 72 hours following oocyte retrieval
  The proportion of prescribed Tylenol with Codeine (Tylenol #3) utilized 72 hours postoperatively will be assessed by telephone encounter. A total of 10 tablets of Tylenol #3 will be prescribed to each participant. Fewer Tylenol #3 used at the end of this time frame would indicate better outcome.

SECONDARY OUTCOMES:
Pain score in post-anesthesia care unit using the Visual Analog Scale | 1-hour after oocyte retrieval
  The Visual Analog Scale will be used to assess postoperative pain 1-hour after egg retrieval. The scale will be in a range from 0 to 10, with 0 being no pain and 10 being unbearable pain. A lower score would indicate a better outcome.
24-hour pain score using the Visual Analog Scale | 24 hours after oocyte retrieval
  The Visual Analog Scale will be used to assess pain 24 hours after egg retrieval. The scale will be in a range from 0 to 10, with 0 being no pain and 10 being unbearable pain. A lower score would indicate a better outcome.
48-hour pain score using the Visual Analog Scale measuring pain | 48 hours after oocyte retrieval
  The Visual Analog Scale will be used to assess pain 48 hours after egg retrieval. The scale will be in a range from 0 to 10, with 0 being no pain and 10 being unbearable pain. A lower score would indicate a better outcome.
72-hour pain score using the Visual Analog Scale measuring pain | 72 hours after oocyte retrieval
  The Visual Analog Scale will be used to assess pain 72 hours after egg retrieval. The scale will be in a range from 0 to 10, with 0 being no pain and 10 being unbearable pain. A lower score would indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Imudia, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ditkoff EC, Plumb J, Selick A, Sauer MV. Anesthesia practices in the United States common to in vitro fertilization (IVF) centers. J Assist Reprod Genet. 1997 Mar;14(3):145-7. doi: 10.1007/BF02766130. PMID 9090556
- [Background] Fiebai PO, Ogunmokun AA, Ajayi RA. Experience with conscious sedation for oocyte retrieval in Nigeria. Afr J Reprod Health. 2008 Apr;12(1):30-4. PMID 20695152
- [Background] Singhal H, Premkumar PS, Chandy A, Kunjummen AT, Kamath MS. Patient Experience with Conscious Sedation as a Method of Pain Relief for Transvaginal Oocyte Retrieval: A Cross Sectional Study. J Hum Reprod Sci. 2017 Apr-Jun;10(2):119-123. doi: 10.4103/jhrs.JHRS_113_16. PMID 28904501
- [Background] Gejervall AL, Stener-Victorin E, Moller A, Janson PO, Werner C, Bergh C. Electro-acupuncture versus conventional analgesia: a comparison of pain levels during oocyte aspiration and patients' experiences of well-being after surgery. Hum Reprod. 2005 Mar;20(3):728-35. doi: 10.1093/humrep/deh665. Epub 2004 Dec 17. PMID 15608039
- [Background] Ozaltin S, Kumbasar S, Savan K. Evaluation of complications developing during and after transvaginal ultrasound - guided oocyte retrieval. Ginekol Pol. 2018;89(1):1-6. doi: 10.5603/GP.a2018.0001. PMID 29411339
- [Background] Frederiksen Y, Mehlsen MY, Matthiesen SM, Zachariae R, Ingerslev HJ. Predictors of pain during oocyte retrieval. J Psychosom Obstet Gynaecol. 2017 Mar;38(1):21-29. doi: 10.1080/0167482X.2016.1235558. Epub 2016 Sep 27. PMID 27670651
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] van Hoogdalem E, de Boer AG, Breimer DD. Pharmacokinetics of rectal drug administration, Part I. General considerations and clinical applications of centrally acting drugs. Clin Pharmacokinet. 1991 Jul;21(1):11-26. doi: 10.2165/00003088-199121010-00002. PMID 1717195
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324